CLINICAL TRIAL: NCT06625099
Title: Comparison of the Effects of Different Positive Expiratory Pressure Levels on Patient Oxygenation and Mechanical Power Values in Laparoscopic Surgeries
Brief Title: Investigation of the Optimum PEEP Mechanical Power Relationship
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Yuksek, Associate Professor in Anesthesiology, Kocaeli City Hospital
Other Study IDs: 2024-68
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation; Mechanical Power; Optimum PEEP; Laparoscopic Abdominal Surgery
Keywords: Mechanical Power; Optimum PEEP; Laparoscopic abdominal surgery; mechanical Ventilation
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group L: After the study group patients were informed preoperatively and accepted to participate in the study, different mechanical ventilation strategies will be applied to the randomly grouped patients after standard propofol, fentanyl, rocuronium midazolam induction anesthesia according to the groups they are in. Group L patients will be applied standard 5 cmH2O PEEP after anesthesia induction.
  The ventilation parameters and vital signs obtained will be recorded, and the mechanical power applied to the patients will be calculated according to Gattinoni's mechanical power calculation formula in volume controlled patients. The groups will be compared for power hemodynamic values and blood gas for oxygenation.
  Interventions: Other: Mechanical Ventilation (MV) with Low PEEP
- Group O: After the study group patients are informed preoperatively and accepted to participate in the study, different mechanical ventilation strategies will be applied to the patients randomly grouped after standard propofol, fentanyl, rocuronium midazolam induction anesthesia according to their groups. Optimum PEEP will be applied to Group O patients after anesthesia induction, with the highest compliance values.
  The ventilation parameters and vital signs obtained will be recorded and the mechanical power applied to the patients will be calculated according to Gattinoni's mechanical power calculation formula in volume-controlled patients. The groups will be compared in terms of power hemodynamic values and blood gas for oxygenation.
  Interventions: Other: Mechanical Ventilation (MV) with Optimum PEEP

INTERVENTIONS:
Other: Mechanical Ventilation (MV) with Low PEEP — Mechanical Ventilation (MV) with Low PEEP During volume controlled ventilation, blood gas values and mechanical power calculations of patients ventilated at 6-8ml/kg tidal volume and 5cmH2o PEEP, I/E: 1/2, 10-14 frequency ranges will be recorded.
  Groups: Group L
Other: Mechanical Ventilation (MV) with Optimum PEEP — Mechanical Ventilation (MV) with Low PEEP During volume controlled ventilation, blood gas values and mechanical power calculations of patients ventilated at 6-8ml/kg tidal volume and optimum PEEP, I/E: 1/2, 10-14 frequency ranges will be recorded.
  The optimum PEEP will be adjusted by titrating to the highest compliance with the open lung strategy.
  Groups: Group O

SUMMARY:
The aim of this study is to compare the effects of standard and optimum positive end expiratory pressures on mechanical power during laparoscopic surgeries.

DETAILED DESCRIPTION:
Perioperative pulmonary complications and ventilator-associated lung injury are challenging issues for anesthesiologists, especially after laparoscopic surgeries. An increasing number of studies suggest lung protective ventilation (LPV) strategies in these patients. It is recommended that patients&; driving pressure be kept low during LPV and positive expiratory pressure (PEEP) be applied to keep the lungs open. However, high PEEP values cannot be adequately applied in laparoscopic surgeries to reduce the restrictive peak pressure for LPV. In laparoscopic surgeries, the patients position and increased intra-abdominal pressure create pressure on the lungs. However, when the applied positive pressure ventilation is insufficient in patients, it can cause atelectasis, and when it is excessive, it can cause barotrauma or volutrauma. The threshold values determined for all these possible complications during LPV should be evaluated together.

Gattinoni and colleagues (2016) explained the effect of mechanical ventilation on the lungs through a work/time formula and formulated the energy used during this work. The applied energy is spent on opening the lungs and ventilation, while the excess is consumed due to heat and resistance in the respiratory tract. The unit of this energy can be formulated in a simplified way as joule/second. The mechanical power formula makes it easier to follow by providing a single parameter instead of different threshold values for barotrauma, volutrauma and atelectrauma for the lungs. Studies have shown that applying energy over 12.6 joules is associated with lung damage. On the other hand, the relationship between the optimum mechanical power (MP) value during ventilation and low and high PEEP is not yet fully known.

In laparoscopic surgeries, high PEEP application may help keep the lungs open and increase ventilation, but it may cause higher mechanical power application. In this case, the effect of high PEEP application on ventilation and patient outcomes is unclear.

In this study, PEEP values and mechanical power values applied during ventilation in patients who will be operated under laparoscopic surgery will be monitored observationally and the PEEP/MP relationship will be examined in terms of patient oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* within the appropriate age range
* agreeing to participate in the study
* again receiving lancetesthesia
* volume controlled ventilation
* no known lung disease
* no known coronary artery disease
* ASA class 1-2 patients

Exclusion Criteria:

* . Patients who do not want to be included in the study will not be included
* Patients with intraoperative deep hypotension (mean arterial pressure <50) will be excluded.
* Those who develop intraoperative hypothermia or have other anesthesia complications will be excluded.
* Patients who will not be extubated postoperatively will be excluded from the study.
* Those with neurological diseases or those using psychiatric medications will also be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo laparoscopic cholecystectomy in the operating rooms of Kocaeli City Hospital will constitute the study universe.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
Mechanical power value in optimum PEEP | During the intraoperative period laparoscopic surgery
  The primary aim of this study is to calculate the mechanical power values (in Joule/min) applied during ventilation among the optimum positive expiratory pressure values in patients undergoing laparoscopic surgery are higher than in patients applied low PEEP.

SECONDARY OUTCOMES:
Effect of high mechanical power on oxygenation in blood gases | During the intraoperative period laparoscopic surgery
  The effect of high mechanical power on oxygenation (Po2 in arterial blood gas analysis) in blood gases; to compare the calculated mechanical power values and partial oxygen pressures in perioperative blood gases between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Yuksek, Md, Study Chair — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study patients belong to Kocaeli City Hospital and it is forbidden to share them.

REFERENCES:
- [Background] Jo YY, Chang YJ, Lee D, Kim YB, Jung J, Kwak HJ. Comparisons of Mechanical Power and Respiratory Mechanics in Pressure-Controlled Ventilation and Volume-Controlled Ventilation during Laparoscopic Cholecystectomy in Elderly Patients. J Pers Med. 2023 Jan 23;13(2):201. doi: 10.3390/jpm13020201. PMID 36836435
- [Background] Pozzi T, Coppola S, Catozzi G, Colombo A, Chioccola M, Duscio E, Di Marco F, Chiumello D. Mechanical power during robotic-assisted laparoscopic prostatectomy: an observational study. J Clin Monit Comput. 2024 Oct;38(5):1135-1143. doi: 10.1007/s10877-024-01170-1. Epub 2024 Jun 17. PMID 38884875
- [Background] Romitti F, Busana M, Palumbo MM, Bonifazi M, Giosa L, Vassalli F, Gatta A, Collino F, Steinberg I, Gattarello S, Lazzari S, Palermo P, Nasr A, Gersmann AK, Richter A, Herrmann P, Moerer O, Saager L, Camporota L, Marini JJ, Quintel M, Meissner K, Gattinoni L. Mechanical power thresholds during mechanical ventilation: An experimental study. Physiol Rep. 2022 Mar;10(6):e15225. doi: 10.14814/phy2.15225. PMID 35340133
- [Background] Gattinoni L, Marini JJ, Collino F, Maiolo G, Rapetti F, Tonetti T, Vasques F, Quintel M. The future of mechanical ventilation: lessons from the present and the past. Crit Care. 2017 Jul 12;21(1):183. doi: 10.1186/s13054-017-1750-x. PMID 28701178
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Silva PL, Ball L, Rocco PRM, Pelosi P. Physiological and Pathophysiological Consequences of Mechanical Ventilation. Semin Respir Crit Care Med. 2022 Jun;43(3):321-334. doi: 10.1055/s-0042-1744447. Epub 2022 Apr 19. PMID 35439832
- [Background] Paudel R, Trinkle CA, Waters CM, Robinson LE, Cassity E, Sturgill JL, Broaddus R, Morris PE. Mechanical Power: A New Concept in Mechanical Ventilation. Am J Med Sci. 2021 Dec;362(6):537-545. doi: 10.1016/j.amjms.2021.09.004. Epub 2021 Sep 28. PMID 34597688